CLINICAL TRIAL: NCT00743288
Title: A Phase I/II Study of Oral Melphalan Combined With LBH589 for Patients With Relapsed or Refractory Multiple Myeloma (MM)
Brief Title: Melphalan and Panobinostat (LBH589) for the Treatment of Patients With Recurrent Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000612441; ONCOTHER-CLBH589BUS15T (Other: Oncotherapeutics); LBH (Other: Oncotherapeutics)
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melphalan and Panobinostat (Experimental): Schedule A: 10mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1-4 of a 28-day cycle and melphalan PO at 0.05 mg/kg on days 1-5 of week 1.
  Toxicity led to the following changes in dose and schedule Schedule B1: 10mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1-4 and 0.05 mg/kg melphalan PO on days 1, 3 and 5 of week 1.
  Schedule B2: 20mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1-4 and 0.05 mg/kg melphalan POon days 1, 3 and 5 of week 1.
  Schedule C: 20mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1 and 2 and 0.05 mg/kg melphalan PO on days 1, 3 and 5 of week 1 Schedule D1: 15 mg/daily LBH589 PO and 0.05 mg/kg melphalan PO on days 1, 3 and 5 of week 1.
  Schedule D2: 15 mg/daily LBH589 PO and 0.10 mg/kg melphalan PO on days 1, 3 and 5 of week 1.
  Schedule D3: 20 mg/daily LBH589 PO and 0.05 mg/kg melphalan PO on days 1, 3 and 5 of week 1.
  Interventions: Drug: Melphalan; Drug: Panobinostat

INTERVENTIONS:
Drug: Melphalan — Same as above
  Other Names: Phenylalanine mustard, Alkeran
Drug: Panobinostat
  Other Names: LBH589

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Panobinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving melphalan together with panobinostat may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of melphalan when given together with panobinostat in treating patients with recurrent multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the maximum tolerated dose (MTD) and determine the dose-limiting toxicities (DLT) of panobinostat in combination with melphalan in patients with relapsed or refractory multiple myeloma. (Phase I)
* To determine the dose of this regimen to be used in the Phase II portion of the study. (Phase I)
* To determine the efficacy as evidenced by the response rate (combined complete response, very good partial response, partial response, and minimal response) in patients treated with this regimen. (Phase II)

Secondary

* To obtain preliminary evidence of efficacy of the combination of LBH589 and melphalan for patients with relapsed or refractory multiple myeloma. (Phase I)
* To determine the safety and tolerability of this regimen in these patients. (Phase II)
* To determine time to disease progression, time to response, and duration of response in patients treated with this regimen. (Phase II)
* To determine progression-free survival and overall survival of patients treated with this regimen. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study followed by a phase II study.

Patients receive oral panobinostat once daily on days 1, 3, 5, 8, 10, and 12 and oral melphalan once daily on days 1, 3 and 5. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of multiple myeloma, based on the following criteria:

  * Major criteria

    * Plasmacytomas on tissue biopsy (1)
    * Bone marrow plasmacytosis (> 30% plasma cells) (2)
    * Monoclonal immunoglobulin (Ig) spike on serum electrophoresis, IgG > 3.5 g/dL or IgA > 2.0 g/dL, and kappa or lambda light chain excretion > 1 g/day on 24-hour urine protein electrophoresis (3)
  * Minor Criteria

    * Bone marrow plasmacytosis (10-30% plasma cells) (a)
    * Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria (b)
    * Lytic bone lesions ©)
    * Normal IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL (d)
  * Meets any of the following sets of multiple myeloma diagnostic criteria:

    * Any two of the major criteria
    * Major criterion 1 plus minor criterion b, c, or d
    * Major criterion 3 plus minor criterion a or c
    * Minor criteria a, b, and c, OR a, b, and d
* Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of ≥ 1 g/dL and/or urine monoclonal immunoglobulin spike of ≥ 200 mg/24 hours, or evidence of lytic bone disease
* Must have received ≥ 1 prior treatment regimen OR refractory to most recent chemotherapy

  * Relapsed following stabilization or response to standard first-line chemotherapy (e.g., vincristine, doxorubicin hydrochloride, and prednisone or melphalan and prednisone) or first-line high-dose chemotherapy
  * Refractory (i.e., failure to achieve at least complete or partial response or stable disease) to most recent chemotherapy, whether or not containing systemic corticosteroids
  * Prior treatment with ≤ 4 days of a total of 400 mg of prednisone (or an equivalent potency of another steroid) for myeloma is not considered a regimen
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy > 3 months
* Platelet count ≥ 75 x 10^9/L (≥ 50 x 10^9/L if bone marrow is extensively infiltrated)
* Absolute neutrophil count ≥ 1.5 x 10^9/L (≥ 1.0 x 10^9/L if bone marrow is extensively infiltrated)
* Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 2.5 times upper limit of normal (ULN)
* Serum bilirubin ≤ 1.5 times ULN
* Creatinine clearance ≥ 30 mL/min; creatinine > 10 mL/min and < 30 mL/min due to significant myelomatous involvement of the kidneys allowed with medical director approval
* Serum potassium ≥ lower limit of normal (LLN)
* Serum magnesium ≥ LLN
* Serum phosphorus ≥ LLN
* Prior localized radiotherapy

Exclusion criteria:

* Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes (POEMS syndrome)
* Plasma cell leukemia
* Pregnant or nursing females; fertile patients must use effective contraception
* Peripheral neuropathy > grade 2
* Impaired cardiac function or clinically significant cardiac disease (including congenital long QT syndrome, history or presence of sustained ventricular tachyarrhythmia; history of ventricular fibrillation or Torsade de Pointes; bradycardia, defined as heart rate (HR) < 50 beats per minute (bpm) [pacemaker allowed provided HR ≥ 50 bpm]; corrected QT interval > 450 msec on screening ECG; left ventricular ejection fraction below normal on screening ECHO or multigated acquisition (MUGA) scan; right bundle branch block with left anterior hemiblock (bifascicular block); myocardial infarction or unstable angina within the past 6 months; New York Heart Association class III-IV congestive heart failure; uncontrolled hypertension; history of labile hypertension; history of poor compliance with an antihypertensive regimen)
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat
* Prior malignancy within the past 5 years except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix
* Other concurrent severe and/or uncontrolled medical or psychiatric conditions (e.g., uncontrolled diabetes or active or uncontrolled infection), including abnormal laboratory values that could cause unacceptable safety risks or compromise protocol compliance
* Known positivity for HIV or hepatitis B or C
* Severe hypercalcemia (i.e., serum calcium ≥ 14 mg/dL)
* Significant history of non-compliance to medical regimens or unwillingness or inability to comply with instructions given by the study staff
* Concurrent medication that risk prolonging the QT interval or inducing Torsades de Pointes
* Prior panobinostat
* Received chemotherapy, bortezomib, thalidomide, lenalidomide or arsenic trioxide within 3 wks of enrollment (with the exception of nitrosoureas within 6 wks of enrollment)
* Received corticosteroids (>10 mg/day prednisone or equivalent) within three weeks before enrollment.
* Received immunotherapy within < 8 weeks; antibody within < 4 weeks; or radiation therapy to > 30% of marrow-bearing bone within < 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (4):
- United States (4):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - James R. Berenson MD, Incorporated, West Hollywood, California
  - Rocky Mountain Cancer Centers - Denver Midtown, Denver, Colorado
  - Center for Cancer and Blood Disorders, Bethesda, Maryland

REFERENCES:
- [Result] Berenson JR, Hilger JD, Yellin O, Boccia RV, Matous J, Dressler K, Ghazal HH, Jamshed S, Kingsley EC, Harb WA, Noga SJ, Nassir Y, Swift RA, Vescio R. A phase 1/2 study of oral panobinostat combined with melphalan for patients with relapsed or refractory multiple myeloma. Ann Hematol. 2014 Jan;93(1):89-98. doi: 10.1007/s00277-013-1910-2. Epub 2013 Oct 18. PMID 24135804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multicenter study
Groups:
- Melphalan and Panobinostat Schedule A: 10mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1-4 of a 28-day cycle and melphalan PO at 0.05 mg/kg on days 1-5 of week 1.
- Melphalan and Panobinostat Schedule B1: 10mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1-4 of a 28-day cycle and melphalan PO at 0.05 mg/kg on days 1, 3 and 5 of week 1.
- Melphalan and Panobinostat Schedule B2: 20mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1-4 of a 28-day cycle and melphalan PO at 0.05 mg/kg on days 1, 3 and 5 of week 1.
- Melphalan and Panobinostat Schedule C: 20 mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1 and 2 of a 28-day cycle and melphalan PO at 0.05 mg/kg on days 1, 3 and 5 of week 1.
- Melphalan and Panobinostat Schedule D1: 15 mg/daily of LBH589 PO and melphalan PO at 0.05 mg/kg on days 1, 3 and 5 of weeks 1 of a 28-day cycle
- Melphalan and Panobinostat Schedule D2: 15 mg/daily of LBH589 PO and melphalan PO at 0.10 mg/kg on days 1, 3 and 5 of weeks 1 of a 28-day cycle
- Melphalan and Panobinostat Schedule D3: 20 mg/daily of LBH589 PO and melphalan PO at 0.05 mg/kg on days 1, 3 and 5 of weeks 1 of a 28-day cycle
Period: Overall Study
Arm/Group | Melphalan and Panobinostat Schedule A | Melphalan and Panobinostat Schedule B1 | Melphalan and Panobinostat Schedule B2 | Melphalan and Panobinostat Schedule C | Melphalan and Panobinostat Schedule D1 | Melphalan and Panobinostat Schedule D2 | Melphalan and Panobinostat Schedule D3
Started | 3 | 3 | 6 | 7 | 6 | 6 | 9 (6 subjects were enrolled in phase 1 and 3 subjects were enrolled as part of the phase 2 expansion.)
Completed | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not Completed | 3 | 3 | 5 | 7 | 6 | 5 | 9
Not completed — Adverse Event | 1 | 1 | 2 | 2 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Progressive disease (PD) | 2 | 0 | 1 | 4 | 5 | 3 | 6
Not completed — Worsening of condition (Not PD) | 0 | 2 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Melphalan and Panobinostat (LBH589): Schedule A: 10mg/daily of LBH589 per orem (PO) on days 1, 3 and 5 of weeks 1-4 of a 28-day cycle and melphalan PO at 0.05 mg/kg on days 1-5 of week 1.
  Toxicity led to the following changes in dose and schedule Schedule B1: 10mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1-4 and 0.05 mg/kg melphalan PO on days 1, 3 and 5 of week 1.
  Schedule B2: 20mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1-4 and 0.05 mg/kg melphalan POon days 1, 3 and 5 of week 1.
  Schedule C: 20mg/daily of LBH589 PO on days 1, 3 and 5 of weeks 1 and 2 and 0.05 mg/kg melphalan PO on days 1, 3 and 5 of week 1 Schedule D1: 15 mg/daily LBH589 PO and 0.05 mg/kg melphalan PO on days 1, 3 and 5 of week 1.
  Schedule D2: 15 mg/daily LBH589 PO and 0.10 mg/kg melphalan PO on days 1, 3 and 5 of week 1.
  Schedule D3: 20 mg/daily LBH589 PO and 0.05 mg/kg melphalan PO on days 1, 3 and 5 of week 1.
Arm/Group | Melphalan and Panobinostat (LBH589)
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 65.4 [34.2 to 88.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 32
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 40
Prior regimens [Median (Full Range); unit: number of prior regimens]
  Number of prior regimens | 4 [1 to 16]
  Number of Bortezomib-containing prior regimens | 2 [0 to 9]

OUTCOME MEASURES:

1. Secondary Outcome: Duration of Response
Time Frame: First evidence of PR or better (for overall response) and MR or better (for clinical benefit response) to start of disease progression or death
Population: Only three patients had responses.
Measure: Median (Full Range); unit: months
Groups:
- Melphalan and Panobinostat Schedule B: B1: 10mg/daily LBH589 on days 1, 3 and 5 of weeks 1-4 and 0.05mg/kg melphalan on days 1, 3 and 5 of week 1.
  B2: 20mg/daily LBH589 on days 1, 3 and 5 of weeks 1-4 and 0.05mg/kg melphalan on days 1, 3 and 5 of week 1.
Arm/Group | Melphalan and Panobinostat Schedule B
Number analyzed (Participants) | 3
months | 8.1 [0 to 17.2]

2. Secondary Outcome: Time to Progression
Time Frame: Time from the start of treatment to progressive disease
Population: All cohorts were analyzed
Measure: Median (Full Range); unit: months
Arm/Group | Melphalan and Panobinostat
Number analyzed (Participants) | 40
months | 1.6 [0.6 to 2.7]

3. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Phase 1: to determine the MTD of panobinostat (LBH589) in combination with melphalan to be used in the Phase 2 portion of the study
Time Frame: 12 months
Population: MTD for Melphalan and Panobinostat was reached in the cohort of 6 participants who received 20 mg/daily LBH589 PO and melphalan PO at 0.05 mg/kg on days 1, 3 and 5 of week 1 of each cycle. Three additional patients were enrolled as part of the phase 2 expansion.
Measure: Number; unit: mg LBH589
Groups:
- Melphalan and Panobinostat Schedule D3: 20mg daily LBH589 and 0.05mg/kg melphalan on days 1, 3 and 5 of week 1
Arm/Group | Melphalan and Panobinostat Schedule D3
Number analyzed (Participants) | 6
mg LBH589 | 20

4. Primary Outcome: MTD
Description: Phase 1: to determine MTD of melphalan in combination with panobinostat to be used in the Phase 2 portion of the study
Time Frame: 12 months
Measure: Number; unit: mg/kg melphalan
Arm/Group | Melphalan and Panobinostat Schedule D3
Number analyzed (Participants) | 6
mg/kg melphalan | 0.05

5. Primary Outcome: Overall Response Rate (ORR) and Clinical Benefit Rate (CBR) [ORR= Complete Response (CR) + Very Good Partial Response (VGPR) + Partial Response (PR)]; CBR=ORR + Minimal Response (MR)] Following Treatment With Panobinostat and Melphalan
Description: Responses were evaluated according to criteria modified from those developed by Blade et al., 1998 The reference point for evaluating response improvement is the baseline. This baseline reference point is also valid when a patient has already achieved a response and transitions through into a better response grade.
Time Frame: 24 months
Measure: Number; unit: participants
Groups:
- Melphalan and Panobinostat Schedule B: Schedules B1 and B2 B1: 10 mg/daily LBH589 on days 1, 3 and 5 of weeks 1-4 of a 28 day schedule and 0.04 mg/kg melphalan on days 1, 3 and 5 of week 1.
  B2:20 mg/daily LBH589 on days 1, 3 and 5 of weeks 1-4 of a 28 day schedule and 0.04 mg/kg melphalan on days 1, 3 and 5 of week 1
- Melphalan and Panobinostat Schedule C: 0.05 mg/kg melphalan on days 1, 3 and 5 of week 1 and 20 mg of LBH589 on days 1, 3, and 5 of weeks 1 and 2.
- Melphalan and Panobinostat Schedule D: Schedules D1, D2 and D3
  D1:LBH589 15mg/daily and melphalan 0.05mg/kg on days 1, 3 and 5 of week 1 D2: LBH589 15mg and daily melphalan 0.10 mg/kg on days 1, 3 and 5 of week 1 D3: LBH589 20mg daily and melphalan 0.05mg/kg on days days 1, 3 and 5 of week 1
- Melphalan and Panobinostat All Patients: Data for all patients irrespective of dosage
Arm/Group | Melphalan and Panobinostat Schedule A | Melphalan and Panobinostat Schedule B | Melphalan and Panobinostat Schedule C | Melphalan and Panobinostat Schedule D | Melphalan and Panobinostat All Patients
Number analyzed (Participants) | 3 | 9 | 7 | 21 | 40
participants
  CR | 0 | 0 | 0 | 0 | 0
  VGPR | 0 | 2 | 0 | 0 | 2
  PR | 0 | 1 | 0 | 0 | 1
  MR | 0 | 0 | 0 | 0 | 0
  SD (stable disease) | 1 | 5 | 5 | 12 | 23
  Progressive disease (PD) | 2 | 1 | 2 | 9 | 14
  ORR (CR+VGPR+ PR) | 0 | 3 | 0 | 0 | 3
  CBR (ORR+MR) | 0 | 3 | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Melphalan and Panobinostat
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 22/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan and Panobinostat (N=40)
Vertebral compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Gram-negative sepsis (Infections and infestations) | 1 (1)
Deep vein thrombosis with oulmonary embolism (Vascular disorders) | 1 (1)
Altered mental status (Psychiatric disorders) | 1 (1)
Hypecalcemia (Metabolism and nutrition disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan and Panobinostat (N=40)
Anemia (>=grade 3) (Blood and lymphatic system disorders) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 9 (9)
Neutropenia (Blood and lymphatic system disorders) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No